CLINICAL TRIAL: NCT05948423
Title: Effect of Tissue Flossing Technique in Patients With Post Traumatic Elbow Stiffness.
Brief Title: Tissue Flossing Technique on Post Traumatic Elbow Stiffness.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah IU Maria Ajaz Mughal
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Elbow Stiffness
Keywords: Tissue Flossing, Postoperative elbow stiffness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group A) Tissue Flossing + Conventional Therapy (Experimental): 1. Tissue Flossing (3reps of 6 different active and passive movements, total 1-2 mints)
  2. Hot Pack (10 mints)
  3. PNF technique on Bicep, Tricep, pronator, Supinator muscle (3reps* 26sec, total 6 mints)
  4. Joint Mobilization (3 reps of humeroulnar and radial head mobilization, total 6 mints) Total treatment duration was 24 mints.
  Interventions: Other: Tisue Flossing Technique
- (Group B) Conventional Therapy (Active Comparator): 1. Hot Pack (10 mints)
  2. PNF technique on Bicep, Tricep, pronator, supinator muscle (3reps* 26sec, total 6 mints)
  3. Joint Mobilization (3 reps of humeroulnar and radial head mobilization, total 6 mints)
  Total treatment duration was 24 mints.
  Interventions: Other: Tisue Flossing Technique

INTERVENTIONS:
Other: Tisue Flossing Technique — Experimental Group (Tissue Flossing + conventional therapy) Tissue Flossing involved active and passive movement with elbow wrapped with a floss band made from latex rubber (7m x 2 inch) Floss band was wrapped around the elbow (distal to proximal) using 25% overlapping pattern with an elongation stretch of 25%. During treatment the compression of floss band was measured with modified sphygmomanometer by placing cuff under floss band (which is applied on muscle) and note the pressure on manometer.
  Control Group (Conventional Therapy) Conventional therapy was applied for 23 minutes for both groups which include hot pack for 10 minutes, PNF (hold-relax with agonist contraction): It started with a gentle stretch of bicep muscle for 10 seconds followed by isometric contraction for 6 seconds then the patient tried to flex their elbow and the therapist also assisted.
  Other Names: Conventional Physical therapy

SUMMARY:
The purpose of this research is to determine the effect of tissue flossing technique on post-traumatic elbow stiffness, Pain and ROM. A randomized control trial was conducted at Pakistan ordinance factory (POF) Hospital Wah Cantt, Pakistan. The sample size was 36 calculated from G-power. 6 participants were excluded from the study and remaining 30 participants were divided into two groups, each having 15 participants. The study duration was six months. Sampling technique was applied was Non probability Convenience Sampling technique for recruitment and group randomization using random selection of participants. Both post-traumatic and post-operative male and female participants of aged 18-45 years with flexion <120° and loss of extension >30°. Tools used in this study are Liverpool elbow Score Questionnaire (LES), Goniometer and Visual Analogue Scale (VAS). Data was analyzed through SPSS version 23.

DETAILED DESCRIPTION:
Post traumatic or operative stiffness at elbow is quite common problem causes higher level of impairments in daily living activities i.e. use of mobile or computer, personal hygiene, dressing, eating, cooking that requires higher degree of elbow range of motion and adversely effects the quality of life (1).

The common reason of stiffness in elbow is trauma with rates ranging from 3% to 20% (1). Incidence of (PTES) is increased up to 56% after elbow trauma (2). Simultaneously radial head and elbow injuries increase incidence rate up to 90%, and 5-10% patients are effected by PTES even with an isolated injury to the radial head (3). Another study shows that exact incidence of elbow stiffness is not known but elbow injuries causes stiffness in approximately 12% of patients (1). Elbow stiffness causes can be categorized as traumatic, atraumatic and congenital (4).

Patients with well reduced and stabilized fracture are also suffer for soft tissue and capsule thickening leads to range of motion limitation. Stiff elbow has thickened capsule with high level of myofibroblast. This causes alteration in the auto-regulation of (TGF-β) transforming growth factor-beta. The influence of myofibroblasts is increased in initial period after trauma but deficient in chronic stiffness (>5 months) (4).

Treatment depends upon the cause of stiffness, stiffness time, severity of stiffness and involved movement of elbow (5). Treatment include CPM (continuous Passive motion), manipulation, stretching, active and passive exercises, mobilization, passive resistance exercises, passive mobilization with movements and PNF (proprioceptive neuromuscular facilitation technique) (6, 7). Physiotherapy is commonly used treatment both for prevention of post traumatic elbow stiffness and regain motion after surgery (7). Factors effecting PTES consist of patients and characteristics of fracture and treatment of fracture causes stiffness, pain, instability and functional limitations of elbow (4).

Clinically according to the severity, elbow stiffness is classified as very severe ( flexion/ extension arc <30), severe ( 30-60), moderate ( 61-90), minimal ( >90) (8). Diagnosis depends upon history, imaging and physical examination. Plain radiographs are useful to see joint congruity, osteophytes and myositis mass (6).

Different studies have been conducted to show influence of tissue flossing on ROM, majority of these studies have shown positive effects on range of motion (9).

A systematic and evidence based search of relevant literature was performed by utilizing Google Scholar as Search engine and the Key words used were Elbow stiffness, Tissue Flossing, Post- Operative elbow stiffness. The purpose of the Literature review is to find out the pre-existing literature regarding the Tissue flossing effects.

In 2017 kiefer et al, conducted a pilot study on the tissue flossing effects and glenohumeral flexibility and concluded that flexibility in posttest is significantly increased (10).

In 2020 Kaneda et al. conducted an experimental research on tissue flossing effect and stretching on calf muscles in which 20 healthy young men participated and concluded that prep and post changes in dorsiflexion was significantly increase with flossing compare to rest (11).

Although enough researches have not been conducted in disease population but some studies have shown its beneficial effect in reducing pain and improve range of motion in diseases population (12, 13).

In 2017, Borda and Selhorst conducted a case study on 14 years old female with chronic pain with 8/10 intensity of Achilles tendinopathy and only two session with tissue flossing shows improvement in pain with 0/10 and disability during sports (12).

In 2018, weber et al. conducted a study on 14 years old male soccer player with Osgood-Schlatter's disease and concluded that there is significant improvement on muscle functions and pain with nine weeks flossing intervention plan (13).

In 2020 by Marco et al. a pilot study was conducted on five young male athletes with knee pain and shows significant improvement on knee pain and jump performance with flossing technique (14).

In 2017 a research was conducted on twelve elite healthy tennis players in which floss band wrapped with 50% stretch on elbow joint and perform 6 passive exercises in three mints and concluded that there is significant improvement in elbow range of motion in floss band group (15).

In 2019, Stevenson conducted a research on 5 male athletes who had stiffness, tightness, heel pain or calf pain and concluded that there was a significant difference between floss group and control group (16).

In 2020, Kielur and powden perform systematic review and meta-analysis in which 6 articles were enrolled and concluded that floss band is an effective method for endurance, strength and physical functions (17)

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18-45 years
* Both male and female
* Complete bone healing
* Immobilization period 4-10 weeks
* Flexion <120° and loss of extension >30°

Exclusion Criteria:

* Those patient who have allergy to latex
* Skin diseases
* Venous Thrombotic disease
* Cardio Pulmonary illness with Grade 3and 4
* Myositis Ossificance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Liverpool Elbow Scoring Questionnaire (LES) | 6 months
  Liverpool elbow Score is valid questionnaire specifically used to assess the functional scoring of elbow joint in elbow stiffness patients. LES contains nine-item (PAQ, P1-P9) patient-answered questionnaire along with six-item (CAS, C1-C6) clinical assessment score. All PAQ and CAS items were calculated with 0 to 10 numbers scale in which the lesser scores denoted greater symptom and functional severity. This scale has Good-to-excellent validity (0.45-0.89) (23).
Goniometer | 6 months
  Universal goniometer measurements at Elbow ROM. The reliability ranged from 0.93 to 0.98 for the goniometric measurements (19).
Visual Analogue Scale | 6 months
  Pain intensity of elbow was measured by using Visual Analogue scale (VAS). VAS is mostly used assessment tool for intensity of pain in rehabilitation. It consists of unmarked 10cm horizontal line in which a patient mark on the line the point that they feel represents the perception of their pain ranges from '0cm' no pain to '100cm' very severe pain. The validity of VAS is 0.7 and reliability is (0.5) (48).

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScNMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Ordinance Factory Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The data will be treat confidentially and only use for the study purpose

REFERENCES:
- [Background] Gracitelli MEC, Guglielmetti CLB, Botelho CAS, Malavolta EA, Assuncao JH, Ferreira Neto AA. Surgical Treatment of Post-traumatic Elbow Stiffness by Wide Posterior Approach. Rev Bras Ortop (Sao Paulo). 2020 Oct;55(5):570-578. doi: 10.1055/s-0039-1700827. Epub 2020 Jan 9. PMID 33093721
- [Background] Liu W, Sun Z, Xiong H, Liu J, Lu J, Cai B, Wang W, Fan C. What are the prevalence of and factors independently associated with depression and anxiety among patients with posttraumatic elbow stiffness? A cross-sectional, multicenter study. J Shoulder Elbow Surg. 2022 Mar;31(3):469-480. doi: 10.1016/j.jse.2021.11.014. Epub 2021 Dec 27. PMID 34968692
- [Background] Englert C, Zellner J, Koller M, Nerlich M, Lenich A. Elbow dislocations: a review ranging from soft tissue injuries to complex elbow fracture dislocations. Adv Orthop. 2013;2013:951397. doi: 10.1155/2013/951397. Epub 2013 Oct 21. PMID 24228180
- [Background] Masci G, Cazzato G, Milano G, Ciolli G, Malerba G, Perisano C, Greco T, Osvaldo P, Maccauro G, Liuzza F. The stiff elbow: Current concepts. Orthop Rev (Pavia). 2020 Jun 25;12(Suppl 1):8661. doi: 10.4081/or.2020.8661. eCollection 2020 Jun 29. PMID 32913596
- [Background] Ritali A, Rotini R, Cavallo M, Marinelli A, Guerra EJLS-J. Instability/stiffness in elbow fracture dislocation. 2020;34:30-5.
- [Background] Mittal R. Posttraumatic stiff elbow. Indian J Orthop. 2017 Jan-Feb;51(1):4-13. doi: 10.4103/0019-5413.197514. PMID 28216745
- [Background] Zhang D, Nazarian A, Rodriguez EK. Post-traumatic elbow stiffness: Pathogenesis and current treatments. Shoulder Elbow. 2020 Feb;12(1):38-45. doi: 10.1177/1758573218793903. Epub 2018 Aug 8. PMID 32010232
- [Background] Marinelli A, Bettelli G, Guerra E, Nigrisoli M, Rotini R. Mobilization brace in post-traumatic elbow stiffness. Musculoskelet Surg. 2010 May;94 Suppl 1:S37-45. doi: 10.1007/s12306-010-0068-5. PMID 20383680
- [Background] Konrad A, Mocnik R, Nakamura M. Effects of Tissue Flossing on the Healthy and Impaired Musculoskeletal System: A Scoping Review. Front Physiol. 2021 May 21;12:666129. doi: 10.3389/fphys.2021.666129. eCollection 2021. PMID 34093228
- [Background] Kiefer BN, Lemarr KE, Enriquez CC, Tivener KA, Daniel TJIJoAT, Training. A pilot study: perceptual effects of the voodoo floss band on glenohumeral flexibility. 2017;22(4):29-33.
- [Background] Kaneda H, Takahira N, Tsuda K, Tozaki K, Sakai K, Kudo S, et al. The effects of tissue flossing and static stretching on gastrocnemius exertion and flexibility. 2020;28(2):205-13.
- [Background] Borda J, Selhorst M. The use of compression tack and flossing along with lacrosse ball massage to treat chronic Achilles tendinopathy in an adolescent athlete: a case report. J Man Manip Ther. 2017 Feb;25(1):57-61. doi: 10.1080/10669817.2016.1159403. Epub 2016 May 30. PMID 28855793
- [Background] Weber PJJoB, Therapies M. Flossing: An alternative treatment approach to Osgood-Schlatter's disease: Case report of an adolescent soccer player. 2018;22(4):860-1.
- [Background] . García-Luna MA, Cortell-Tormo JM, González-Martínez J, García-Jaén M. The effects of tissue flossing on perceived knee pain and jump performance: A pilot study. 2020.
- [Background] Hodeaux K. The effect of floss bands on elbow range of motion in tennis players: University of Arkansas; 2017.
- [Background] Stevenson P, Stevenson R, Duarte KWJJMBAS. Acute effects of the voodoo flossing band on ankle range of motion. 2019;7(6):244-53.
- [Background] Kielur DS, Powden CJ. Changes of Ankle Dorsiflexion Using Compression Tissue Flossing: A Systematic Review and Meta-Analysis. J Sport Rehabil. 2020 Oct 19;30(2):306-314. doi: 10.1123/jsr.2020-0129. PMID 33075750
- [Background] Wilson RC, Jones PW. A comparison of the visual analogue scale and modified Borg scale for the measurement of dyspnoea during exercise. Clin Sci (Lond). 1989 Mar;76(3):277-82. doi: 10.1042/cs0760277. PMID 2924519
- [Background] Sun Z, Fan C. Validation of the Liverpool Elbow Score for evaluation of elbow stiffness. BMC Musculoskelet Disord. 2018 Aug 21;19(1):302. doi: 10.1186/s12891-018-2226-0. PMID 30126385